CLINICAL TRIAL: NCT02932488
Title: Cerebral Pharmacodynamic Effects of 5-HT1B Receptor Stimulation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pilot study with sumatriptan found no significant changes in the primary outcome parameter (change in CBF)
Sponsor: Gitte Moos Knudsen (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Chair, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NP3
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
Keywords: PET-MR; 5-HT1B receptor; Sumatriptan; phMRI; [11C]AZ10419369
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sumatriptan (Experimental): In the pilot study (an MR-only study) subjects will receive up to five doses of sumatriptan in the range of 10 ug/kg to 80 ug/kg. This allows us to establish a dose-response curve for each subject. Administration of sumatriptan in the pilot study will be spaced with approximately one week apart to avoid carry-over effects of the drug.
  In the main study (a PET-MR study), the sumatriptan dose with the maximal effect size and minimum side effects will be used for all subjects.
  Interventions: Drug: Sumatriptan

INTERVENTIONS:
Drug: Sumatriptan — Sumatriptan is a 5-HT1B receptor agonist used for treatment of migraine attacks
  Other Names: Imigran

SUMMARY:
The purpose of this study is to show that PET-MR imaging can be used for obtaining a pharmacodynamic profile of drugs. By using the 5-HT1B receptor as target we also aim to find effect areas and sizes of the 5-HT1B receptor agonist sumatriptan.

DETAILED DESCRIPTION:
Recent technological advances in multimodal imaging have enabled the simultaneous acquisition of magnetic resonance imaging (MRI) and PET data. Whereas functional MRI (fMRI) provides excellent spatio-temporal resolution for localizing changes in brain activity, PET offers high sensitivity and neurochemical specificity. Together, PET and MRI measures have the potential to help clarify the neurochemical basis of changes in fMRI signal induced by selective exogenous ligands or endogenous neurotransmitter.

In the present study we will target the 5-HT1B receptor for which a selective radioligand exist (11C-AZ10419369). The receptor can be stimulated with the agonist sumatriptan, which is used for alleviating migraine attacks. The mechanism of action of sumatriptan is not precisely known and it is unknown to what degree sumatriptan crosses the blood-brain barrier and exerts its effect in the parenchyma. In this study we can determine the blood brain barrier penetration of sumatriptan and thereby evaluate Effect sizes, distribution of signal changes, and correlation between the occupancy at the 5-HT1B receptor in the parenchyma (measured by changes in BPND) and the hemodynamic response (measured by changes in CBF).

Ahead of the main study a pilot study will be conducted in which increasing doses of sumatriptan will be tested in the same subject to obtain a dose-response curve. At the same time side effects will be observed and scored. This serves to find the dose with maximum effect size but minimal side effects, which can then be used in the main study for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age 18-60

Exclusion Criteria:

* Primary psychiatric disease (DSM IV Axis I or WHO ICD-10 diagnostic classification).
* Present or former neurological diseases,
* Severe somatic disease
* Medication that can interfere with the test results.
* Doesn't speak Danish fluently or is severely, visually or hearing impaired.
* Information regarding former learning disabilities.
* Pregnancy at the time of the scanning
* Breast feeding
* MR-scanner incompatibility (metal in soft tissue)
* Alcohol or drug abuse
* Allergy to ingredients in used drugs
* Participation in experiments with radioactivity (>10 mSv) within the last year or considerable work-related exposure to radioactivity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Changes in 5-HT1B receptor binding as measured with [11C]AZ10419369 | Two binding potentials are obtained from the 120 min scan: Baseline BPND is determined from 0-50 min. Intervention BPND is determined from 50-120 min.
  Both measures of receptor binding will be calculated from the same PET-MR acquisition.
Changes in cerebral blood flow measured with pseudo continuous Arterial Spin Labeling | CBF is measured 15 min prior and 30 min after the injection of sumatriptan giving 45 min of total CBF measurement time.
  CBF will be measured continuous and within the acquisition a dynamic change in CBF upon administration of sumatriptan will be obtained.

SECONDARY OUTCOMES:
Change in [11C]AZ10419369 concentration in blood and plasma | At 2.5, 20, 49, 51, 90 and 120 min after injection of [11C]AZ10419369
  Blood samples will be drawn throughout the acquisition time and radioactivity in blood and plasma will be measured.
Plasma concentration of sumatriptan | At -1, 1, 10, 20, 35 and 75 min after injection of sumatriptan
  Blood samples will taken to measure the plasma concentration of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, MD, DMSc, Study Chair — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage) data will be available for neuroscience research community contingent on approval by scientific board.